CLINICAL TRIAL: NCT04425967
Title: Short Course Of Preoperative Radiotherapy in Head and Neck-, Trunk- and Extremity Soft Tissue Sarcomas; a Randomized Phase II Clinical Trial
Brief Title: Short Course Of Preoperative Radiotherapy in Head and Neck-, Trunk- and Extremity Soft Tissue Sarcomas
Acronym: SCOPES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20SCP
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcomas
Keywords: preoperative radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: randomization between the standard arm A of 50 Gy in 5 weeks or arm B with hypofractination of 14x3Gy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25x2Gy (Active Comparator): the conventional schedule of 25 x 2 Gy, once daily fractionation in a five-week OTT
  Interventions: Radiation: pre-operative radiotherapy
- 14x3Gy (Experimental): the study schedule of 14 x 3 Gy, once daily fractionation in a three-week overall treatment time
  Interventions: Radiation: pre-operative radiotherapy

INTERVENTIONS:
Radiation: pre-operative radiotherapy — pre-operative radiotherapy
  Other Names: radiotherapy

SUMMARY:
Currently, soft tissue sarcomas (STS) are preoperatively irradiated in a conventionally fractionated regimen of 25 x 2 Gy in five weeks. Recent radiobiological investigations, however, suggest sensitivity to (modest) hypofractionation. Within this study, patients will be randomized to receive either the conventional schedule of 25 x 2 Gy or a shorter preoperative regimen of 14 x 3 Gy, in the hypothesis that both the postoperative wound complication rate until 30 days after surgery, as well as the local control probability at two years are comparable in both arms.

DETAILED DESCRIPTION:
Surgery is the cornerstone in the treatment of non-metastatic sarcomas. Whenever feasible the resection should include a free surgical margin providing a rim of uninvolved tissue surrounding the tumor. In most deep located tumors however, to preserve essential neurovascular and bone structures and thus to preserve function, the margins are often limited. High grade tumors are, even with wider margins, at higher risk of local failure. Radiotherapy can reduce this risk of local failure.

Preoperative radiotherapy does increase the risk for early complications due to unavoidable irradiation of the normal tissues surrounding the sarcoma mass, particularly for lower extremity lesions (6-9).

Preoperative radiotherapy aims to reduce tumor vitality prior to resection, theoretically allowing more conservative surgical therapy. Postoperative RT allows histological examination of the tumor specimen, especially the margins, aiding in further treatment planning; it may also be associated with fewer early wound complications. (10, 11).

In preoperative radiotherapy, as compared to postoperative radiotherapy, lower doses (50 versus 60 to 66 Gy) and smaller field sizes can be used, resulting in a reduced risk of late, often irreversible, complications. Consequently, preoperative RT is the preferred approach in many centers. Although the outcomes of combined RT and surgery are favorable, approximately 15% of the patients may relapse locally and about 30-50% distantly (dependent upon, among others, age, histopathology, size and grade), stressing the need for further improvement. These improvements should not only be sought in the domain of oncological endpoints, but also in decreasing treatment burden. A reduction in treatment duration, maintaining local control rates without increasing the rates of postoperative wound complications would serve the latter endpoints. For this purpose, quality of life questionnaires as well as patient reported outcomes measurements could come of help.Modern radiobiological investigations suggest that, on average, intermediate to high-grade soft tissue sarcomas may have α/β ratio's substantially below 10 Gy, justifying clinical studies exploring the possibility of (modest) hypofractionation. Obviously, various subtype derived cell lines exhibit different characteristics but on average an α/β ratio of 5 Gy would be a reasonable denominator for sarcomas as a group. However, it is important not to exaggerate hypofractionation in a setting where patients still need to undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed intermediate to high grade soft tissue sarcoma localized to the extremities, trunk and chest wall or the head and neck area, for which the standard treatment is a combination of and radiotherapy and surgery (deep seated and/or > 5cm in largest tumor diameter and/or an anticipated close resection margin and/or grade II/III according to the FNCLCC definition);
* • Absence of regional and/or distant disease. Patients staged by at least a CT scan of the chest (. Staging may also be performed by FDG-PET scanning and or total body MRI scans. Patients with an uncertain metastatic status (e.g. small indifferent lung nodules) and patients with a low metastatic burden not precluding the application of both preoperative radiotherapy and definitive surgery, are allowed to participate;
* WHO Performance Status ≤ 2;
* Able and willing to undergo preoperative radiotherapy;
* Able and willing to undergo definitive surgery;
* Able and willing to comply with regular follow-up visits;
* Able and willing to complete patient reported outcome questionnaires (health-related quality of life and cost effectiveness);

  • Able and willing to undergo randomization;
* Age ≥ 18 years;
* Signed written informed consent

Exclusion Criteria:

* Prior malignancies; except another malignancy and disease-free for ≥ 5 years, or completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma;
* Patients with recurrent sarcomas who underwent prior radiotherapy to the target lesion (if the primary sarcoma was managed by surgery only and no perioperative RT, patients are eligible);
* Ewing sarcoma and other PNET family tumors, rhabdomyosarcomas (both pediatric and adult), osteosarcomas;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Female patients who are pregnant;
* Intention to perform an isolated limb perfusion, instead of a tumor resection;
* Neoadjuvant chemotherapy to be scheduled between end of radiotherapy and definitive surgery (neoadjuvant chemotherapy before radiotherapy is allowed);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
the short-term toxicity | 30 days post operative
  wound complications

SECONDARY OUTCOMES:
local control | During follow up (5 years)
  percentage of patients without local failure after surgery
long-term toxicity | During follow up (5 years)
  fibrosis, edema, joint impairment and bone fractures
Wound complication rate | From surgery until 120 days post-surgery
  the rate of postoperative wound complications between day 31 and day 120 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (4):
- Netherlands (4):
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Radboudumc, Nijmegen
  - Erasmus Medical Centre, Rotterdam

IPD SHARING:
Plan to Share IPD: No